CLINICAL TRIAL: NCT00485706
Title: Arterial Stiffness and Decreased Bone Buffering Capacity in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ML4181; S50455
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Kidney Disease; Hypercalcemia
Keywords: dialysis; vascular calcification; bone mineralism; arterial stiffness; bone metabolism; chronic kidney disease
MeSH Terms: conditions — Kidney Diseases; Hypercalcemia; Vascular Calcification; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: high calcium dialysate

SUMMARY:
Renal patients have an increased risk for cardiovascular complications. There is also increased vascular calcification and bone metabolism is similarly abnormal in patients with chronic kidney disease.

In dialysis patients frequent episodes of hypercalcaemia occur. In a healthy bone structure those episodes of hypercalcemia are buffered by the bone. The absence of bone buffering capacity in dialysis patients can be a mechanism for vascular calcifications.

DETAILED DESCRIPTION:
Study hypothesis.

Patient with a higher ∆ Calcium (Calcium post - Calcium pre) have a diminished bone buffering capacity indicative for adynamic bone disease compared with patients with smaller ∆ Calcium.

This may result in higher extraosseous calcification and higher pulse wave velocity

∆ PTH/∆ Calcium may reflect the sensitivity and density of the calcium receptors; this may reflect parathyroid "health"

ELIGIBILITY:
Inclusion Criteria:

* maintenance hemodialysis patients

Exclusion Criteria:

* dialysis <3 months
* aortobifemoral graft
* calcium level predialysis >10.5 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06

PRIMARY OUTCOMES:
correlation between calcium increase and pulse wave velocity
  correlation between calcium increase and pulse wave velocity
correlation between calcium change and pth change
  correlation between calcium change and pth change

SECONDARY OUTCOMES:
correlation between calcium increase and vascular calcifications
  correlation between calcium increase and vascular calcifications
correlation between calcium change and bone markers
  correlation between calcium change and bone markers

CONTACTS AND LOCATIONS:
Overall Officials: kathleen Claes, MD, Principal Investigator — UZ Gasthuisberg
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium